CLINICAL TRIAL: NCT06370403
Title: Effects of Head and Neck Cooling and Heating on Central and Peripheral Fatigue, Motor Accuracy and Blood Markers of Stress in Multiple Sclerosis and Healthy Men
Brief Title: Effects of Head and Neck Cooling and Heating on Fatigue in Multiple Sclerosis and Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: LithuanianSportsU-21
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis; Cooling; Heating; Fatigue; Exercise
MeSH Terms: conditions — Multiple Sclerosis; Fatigue; Motor Activity

STUDY DESIGN:
Masking Description: The researchers who analyzed the venous blood samples were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cooling of the head and neck in multiple sclerosis and healthy subjects (Experimental): Multiple sclerosis and healthy male subjects participated in the head and neck cooling program. During cooling procedure, the participant performed fatiguing isometric motor task with a head and neck cooling helmet at (18°C next to the head and neck skin).
  Interventions: Other: Cooling of the head and neck
- Heating of the head and neck in multiple sclerosis and healthy subjects (Experimental): Multiple sclerosis and healthy male subjects participated in the head and heating program. During heating procedure, the participant performed fatiguing isometric motor task with a head and neck heating helmet at (43°C± 1°C next to the head and neck skin).
  Interventions: Other: Heating of the head and neck

INTERVENTIONS:
Other: Cooling of the head and neck — Cooling of the head and neck at 18°C next to the head and neck skin in multiple sclerosis and healthy subjects
  Arms: Cooling of the head and neck in multiple sclerosis and healthy subjects
Other: Heating of the head and neck — Heating of the head and neck at 43 ± 1°C next to the head and neck skin in multiple sclerosis
  Arms: Heating of the head and neck in multiple sclerosis and healthy subjects

SUMMARY:
Local head and neck cooling strategies can help reduce multiple sclerosis-related fatigue, while heating can exacerbate heat-related fatigue. However, no study has detailed the peripheral and central responses to head and neck cooling (at 18°C) and heating (at 43 ± 1°C next to the scalp and neck skin) during fatiguing isometric exercise in non-challenging ambient temperature in multiple sclerosis and healthy male subjects. In addition, there is a lack of data describing the effects of head and neck cooling/heating and strenuous exercise on blood markers, muscle temperature, motor accuracy, and rate of perceived exertion. The investigators hypothesized that: (i) men with multiple sclerosis would be more affected by central and peripheral fatigue compared to healthy subjects; (ii) local cooling will result in greater central fatigue but will be associated with greater peripheral fatigue, whereas heating will result in greater central and peripheral fatigue in multiple sclerosis men; (iv) local cooling and heating will have a greater effect on the release of stress hormones, rate of perceived exertion and motor accuracy compared to the control condition in both multiple sclerosis and healthy groups.

ELIGIBILITY:
Inclusion criteria:

* Relapsing-remitting multiple sclerosis disease course according to McDonald criteria
* Expanded Disability Status Scale less than 4 points and Fatigue Severity Scale score greater than 5 points in participants with multiple sclerosis
* Males
* Age between 18 and 45 years
* Sufficient tolerance to electrical stimulation

Exclusion Criteria:

* Physical limitations that would impair the ability to perform neuromuscular testing
* Mental disorders, such as depression or anxiety, due to their recognized association with fatigue
* Involvement in temperature manipulation program for ≥ 3 months
* Attending any excessive physical exercise or sports programs
* With blood/needle phobia

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-02-04 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2017-01-08 (Actual)

PRIMARY OUTCOMES:
Body weight (kg) | Every time in all conditions at the baseline
  Body weight (kg) was evaluated using Tanita Body Composition Analyzer (Japan).
Body fat (%) | Every time in all conditions at the baseline
  Body fat (%) was assessed using Tanita Body Composition Analyzer (Japan).
Body free fat mass (kg) | Every time in all conditions at the baseline
  Body free fat mass (kg) was evaluated using Tanita Body Composition Analyzer (Japan).
Body mass index (kg/m2) | Every time in all conditions at the baseline
  The body mass index (in kg/m2) was defined as the body mass divided by the square of the body height.
Change in muscle temperature (°C) | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  Muscle temperature was measured using a needle microprobe (Intramuscular Probe MKA, thermometer model DM-852, Ellab) inserted approximately 3 cm beneath the skin surface into the vastus lateralis muscle of the right leg.
Change in plasma cortisol (nmol/L) concentrations | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  Plasma cortisol concentrations (nmol/L) were measured using an AIA-2000 automated enzyme immunoassay analyser (Tosoh Corp, Tokyo, Japan).
Change in plasma dopamine (nmol/L) concentrations | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  Dopamine concentrations (nmol/L) were measured using a kit for dopamine enzyme-linked immunosorbent assay (ELISA) (IBL, Hamburg, Germany).
Change in plasma prolactin (ng/mL) concentrations | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  Prolactin levels (ng/mL) were measured using a kit for prolactin ELISA (IBL) and Gemini analyzer (Stratec Biomedical GmbH, Germany).
Change in subjective rating of perceived exertion | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  Perceived exertion was assessed using the Borg scale, ranging from 6 (no exertion) to 20 (maximum exertion).
Change in muscle activity (mV) | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  Vastus medialis and vastus lateralis electromyographic (EMG) amplitude (in mV) parameters of muscular activity were measured using surface EMG (Biometrics, UK) thorough neuromuscular function assessment.
Change in muscle activity (Hz) | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  Vastus medialis and vastus lateralis muscles electromyographic (EMG) frequency (in Hz) parameters of muscular activity were measured using surface EMG (Biometrics, UK) thorough neuromuscular function assessment.
Change in voluntary torque (Nm) | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  Isometric and isokinetic voluntary torques (in Nm) of the quadriceps muscles were measured using an isokinetic dynamometer (Biodex Medical Systems, USA).
Change in involuntary torque (Nm) | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  Involuntary torque of the quadriceps muscles were measured using an isokinetic dynamometer (Biodex Medical Systems, USA) and a high-voltage stimulator (Digitimer DS7A, Digitimer, UK). Peak torques (in Nm) induced by electrical stimulation at 20 Hz,at 100 Hz, and at TT100 were measured.
Change in muscle contraction and relaxation (ms) | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  The contraction and half-relaxation time (in ms) were measured in 100Hz stimulated contractions.
Change in central activation ratio (percent) | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  To evaluate central activation ratio (CAR), a TT-100 Hz stimuli was superimposed on the maximal voluntary contraction (MVC), and the CAR was computed using the following equation: CAR = MVC/(MVC+TT-100 Hz) × 100percent, where where a CAR of 100 percent indicates complete activation of the exercising muscle and a CAR < 100 percent indicates central activation failure or inhibition.
Change in constant error | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  The accuracy of the intermittent isometric contraction tasks was calculated as a constant error. Constant error = ∑(xi - T)/n where xi is the motor task performed (N·m); T is the target quantity, i.e., the motor task required; n is the number of trials; and Σ indicates the mean that was calculated considering the algebraic symbols (±).
Change in absolute error | Baseline, up to 60 minutes, up to 120 minutes, after 180minutes
  The absolute error specifies the absolute deviation from the required target force. Absolute error = ∑|xi - T|/n where xi is the motor task performed (N·m); T is the target quantity, i.e., the motor task required; n is the number of trials; and vertical brackets Σ | | indicate the mean that was calculated without considering the algebraic symbols (±).

SECONDARY OUTCOMES:
Height (m) | Every time in all conditions at the baseline
  Height (in m) was measured using a Harpenden anthropometer set (Holtain Ltd, UK)

CONTACTS AND LOCATIONS:
Overall Officials: Gintarė Daukšaitė, Principal Investigator — Lithuanian Sports University
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania